CLINICAL TRIAL: NCT00075660
Title: A Phase II Study of Triapine (NSC 663249) in Previously Untreated Patients With Recurrent Renal Cell Carcinoma
Brief Title: 3-AP in Treating Patients With Previously Untreated Locally Recurrent or Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I161; CAN-NCIC-IND161 (Other: PDQ); CDR0000347409 (Other: PDQ)
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: triapine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as 3-AP, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of 3-AP in treating patients who have locally recurrent or metastatic renal cell (kidney) carcinoma (cancer).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of 3-AP (Triapine®), in terms of objective response rate, in patients with previously untreated locally recurrent or metastatic renal cell carcinoma.

Secondary

* Determine the adverse events and tolerability of this drug in these patients.
* Determine the time to disease progression and overall survival of patients treated with this drug.

OUTLINE: This is a nonrandomized, multicenter study.

Patients receive 3-AP (Triapine®) IV over 2 hours on days 1-4 and 15-18. Treatment repeats every 28 days for up to 6 courses (for stable patients) in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) receive 1 additional course after documentation of CR. Patients who achieve a partial response (PR) receive 2 additional courses after documentation of stable PR.

Patients are followed every 4 weeks until relapse and then every 3 months for up to 2 years.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed renal cell carcinoma

  * Locally recurrent OR metastatic disease
  * Incurable by standard therapy
* Clinically and/or radiologically measurable disease

  * At least 1 unidimensionally measurable lesion* at least 20 mm by x-ray, physical exam, or non-spiral CT scan OR at least 10 mm by spiral CT scan
  * If the sole site of measurable disease is in a previously irradiated field, there must be documented disease progression at that site NOTE: *Bone lesions are not considered measurable disease
* No documented brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No glucose-6-phosphate dehydrogenase (G6PD) deficiency* NOTE: *Screening for G6PD deficiency is required for patients of African, Asian, or Mediterranean descent

Hepatic

* Bilirubin normal
* AST or ALT no greater than 2.5 times upper limit of normal (ULN)

Renal

* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 50 mL/min

Cardiovascular

* No myocardial infarction within the past 6 months
* No symptomatic congestive heart failure
* No unstable angina
* No active cardiomyopathy
* No cardiac arrhythmia
* No uncontrolled hypertension

Pulmonary

* No pulmonary disease requiring oxygen

Immunologic

* HIV negative
* No known hypersensitivity to compounds of similar chemical or biological composition to 3-AP (Triapine®)
* No active uncontrolled or serious infection
* No immunodeficiency

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other prior malignancy except adequately treated nonmelanoma skin cancer, curatively treated carcinoma in situ of the cervix, or other curatively treated solid tumor with no evidence of disease for at least 5 years
* No history of significant neurologic or psychiatric disorder (e.g., uncontrolled psychotic disorders) that would preclude giving informed consent or complying with study requirements
* No active peptic ulcer disease
* No other serious illness or medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 3 months since prior interferon for advanced or recurrent disease
* No other prior immunotherapy for advanced or recurrent disease
* No prior gene therapy

Chemotherapy

* No prior systemic chemotherapy for advanced or recurrent disease

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy (except low-dose nonmyelosuppressive radiotherapy) and recovered

Surgery

* At least 2 weeks since prior major surgery

Other

* No prior investigational anticancer agents
* No other concurrent anticancer agents or therapy
* No other concurrent investigational therapy
* No concurrent anticoagulants

  * Concurrent nontherapeutic warfarin or heparin allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-05-11 (Actual); Primary Completion 2005-10-04 (Actual); Study Completion 2008-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knox, MD, Study Chair — Toronto General Hospital
Locations (8):
- Canada (8):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Knox JJ, Hotte SJ, Kollmannsberger C, Winquist E, Fisher B, Eisenhauer EA. Phase II study of Triapine in patients with metastatic renal cell carcinoma: a trial of the National Cancer Institute of Canada Clinical Trials Group (NCIC IND.161). Invest New Drugs. 2007 Oct;25(5):471-7. doi: 10.1007/s10637-007-9044-9. Epub 2007 Mar 28. PMID 17393073